CLINICAL TRIAL: NCT02854098
Title: The Comorbidity of Benign Hypermobility Joint Syndrome and Functional Constipation in Children
Acronym: MobCon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Andrzej Załęski, M.D., Medical University of Warsaw
Other Study IDs: 1W33
Record Dates: First submitted 2016-07-16; First posted 2016-08-03 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Benign Hypermobility Syndrome; Functional Constipation
Keywords: BHJS, constipation
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Constipation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- with functional constipation: n = 200 patients with functional constipation examined for BHJS age 3 -18 years meet inclusion criteria, do not fulfill exclusion criteria
- without functional constipation: n = 200 patient with functional constipation examined for BHJS age 3 -18 years meet inclusion criteria, do not fulfill exclusion criteria

SUMMARY:
Benign Hypermobility Joint Syndrome is a group of inherited abnormalities in the structure of connective tissues, manifested by disturbances in the proportion of collagen. The main symptoms of this syndrome include: laxity of joint capsules and ligaments, hypermobility of the joints, as well as numerous disturbances in the functioning of internal organs that contain connective tissue, including the gastrointestinal tract. Hypermobility of joints affects approximately 10% of the population of Western countries, is more common in small children and female. Modified Beighton scale is the basic scale for assessing hypermobility of joints. The scale (as assessed using the goniometer) is a reliable tool for the evaluation of excessive laxity of the connective tissue in children.

Functional constipation is a very common condition, affecting approximately 3-5% of children and adolescents, with peak onset between 2 and 4 years of age. The etiology of this disorder is multifactorial, and till day it is still exactly unknown why some children develop constipation, while in others we can observe the correct scheme of defecation. Suspending stool enhances the retention of fecal masses, which subsequently causes painful defecation. Diagnosis is based on history, clinical symptoms and physical examination. Increased susceptibility of the wall of the distal gastrointestinal tract could explain the predisposition of some children to retain fecal masses and the development of constipation.

Due to the unclear etiology of functional constipation, it seems reasonable to conduct a study assessing whether excessive laxity of connective tissue (assessed on the basis of the hypermobility of the joints) facilitates the accumulation of stool in the large intestine, and so is the one of the reasons leading to development of functional constipation in children.

DETAILED DESCRIPTION:
Clinical question: Is there among patients with functional constipation increased percentage of children with Benign Hypermobility Joint Syndrome, compared with a population of healthy children? In discussion we would like to determine whether the excessive laxity of connective tissue can promote the development of functional constipation in children.

Description of the study:

1. Anamnesis and physical examination of the patient
2. The consent of the parents and the patient (if > 15 years) to participate in the study
3. Determining whether the patient meets the criteria for inclusion in the study
4. The exclusion of patients meeting the exclusion criteria for the study - on the basis of anamnesis and physical examination (including neurological) and diagnostic tests (biochemical and electrolyte TSH -, Na, K, Ca, P, Mg), if indicated
5. In patients classified to the study, the degree of laxity of the connective tissue will be assessed in the basis of modified Beighton scale
6. In the control group - patients without constipation in an interview - the degree of laxity of the connective tissue will be assessed in the basis of modified Beighton scale
7. Evaluation of the results.

Rome III Criteria Functional Constipation

Diagnostic criteria must include one month in children up to 4 years of age and two months in older children(with insufficient criteria for diagnosis of IBS) of at least two of the following:

1. Two or fewer defecations per week
2. At least one episode/week of incontinence after the acquisition of toileting skills
3. History of excessive stool retention
4. History of painful or hard bowel movements
5. Presence of a large fecal mass in the rectum
6. History of large diameter stools which may obstruct the toilet Accompanying symptoms may include irritability, decreased appetite, and/or early satiety. The accompanying symptoms disappear immediately following passage of a large stool.

Modified Beighton scale Hypermobility of joints indicates ≥ 4 points out of 9 possible.

The Beighton score is measured by adding 1 point for each of the following:

1. Placing flat hands on the floor with straight legs
2. Left knee bending backward (>10 °)
3. Right knee bending backward (>10 °)
4. Left elbow bending backward (>10 °)
5. Right elbow bending backward (>10 °)
6. Left thumb touching the forearm
7. Right thumb touching the forearm
8. Left little finger bending backward (>90 °)
9. Right little finger bending backward (>90 °)

ELIGIBILITY:
First group:

Inclusion Criteria:

1. Age 3 - 18 years.
2. Diagnosed functional constipation (on the basis of III Rome Criteria)
3. Informed consent of patients (if more than 16 years) and caregivers

Exclusion Criteria:

1. Organic causes of constipation (anatomical abnormalities: narrowing of the anus or rectum, state after surgical correction of this anomalies)
2. Metabolic and gastrological diseases in anamnesis: hypothyroidism, hypercalcemia, hypokalemia, cystic fibrosis, diabetes, celiac disease
3. Neuropathies: defects and injures of the spinal cord, encephalopathies
4. Neuromuscular disorders: Hirschsprung's disease, intestinal neuronal dysplasia, visceral myopathies and neuropathies
5. Abnormal abdominal musculature: Down syndrome;
6. The use of drugs (opioids, phenobarbital, sucralfate, antidepressants, anticholinergic, sympathomimetic)
7. Lack of informed consent of patients (if more than 16 years) and caregivers

Second group:

Inclusion Criteria:

1. Age 3 - 18 years.
2. Without functional constipation
3. Informed consent of patients and caregivers

Exclusion Criteria:

1 Lack of informed consent of patients and caregivers

Place: Department of Pediatric Gastroenterology and Nutrition, Medical University of Warsaw, Poland

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 2 groups, n = 400 (200 patients each group) age 3 - 18 years. first group - with functional constipation second group - without functional constipation
  Each patient meet inclusion criteria, do not fulfill exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The comorbidity of benign hypermobility joint syndrome and functional constipation in children (in %) | April 2017
  The Hypermobility of the connective tissue as one of the etiological factors of functional constipation in children

SECONDARY OUTCOMES:
The comorbidity of BHJS and functional constipation, depending on age (in %) | April 2017
The comorbidity of BHJS and functional constipation, depending on gender (in %) | April 2017

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Albrecht, PhD, Study Chair — Department of Pediatric Gastroenterology and Nutrition, Medical University of Warsaw
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mirska A, Kalinowska AK, Topór E, et al. Łagodny zespół hipermobilności stawów (BHJS). Neurologia Dziecięca 2011; 41; 135-140.
- [Background] Kovacic K, Chelimsky TC, Sood MR, Simpson P, Nugent M, Chelimsky G. Joint hypermobility: a common association with complex functional gastrointestinal disorders. J Pediatr. 2014 Nov;165(5):973-8. doi: 10.1016/j.jpeds.2014.07.021. Epub 2014 Aug 20. PMID 25151198
- [Background] Fikree A, Grahame R, Aktar R, Farmer AD, Hakim AJ, Morris JK, Knowles CH, Aziz Q. A prospective evaluation of undiagnosed joint hypermobility syndrome in patients with gastrointestinal symptoms. Clin Gastroenterol Hepatol. 2014 Oct;12(10):1680-87.e2. doi: 10.1016/j.cgh.2014.01.014. Epub 2014 Jan 16. PMID 24440216
- [Background] Grahame R, Bird HA, Child A. The revised (Brighton 1998) criteria for the diagnosis of benign joint hypermobility syndrome (BJHS). J Rheumatol. 2000 Jul;27(7):1777-9. No abstract available. PMID 10914867
- [Background] Smits-Engelsman B, Klerks M, Kirby A. Beighton score: a valid measure for generalized hypermobility in children. J Pediatr. 2011 Jan;158(1):119-23, 123.e1-4. doi: 10.1016/j.jpeds.2010.07.021. Epub 2010 Sep 17. PMID 20850761
- [Background] Zarate N, Farmer AD, Grahame R, Mohammed SD, Knowles CH, Scott SM, Aziz Q. Unexplained gastrointestinal symptoms and joint hypermobility: is connective tissue the missing link? Neurogastroenterol Motil. 2010 Mar;22(3):252-e78. doi: 10.1111/j.1365-2982.2009.01421.x. Epub 2009 Oct 15. PMID 19840271
- [Background] Mohammed SD, Lunniss PJ, Zarate N, Farmer AD, Grahame R, Aziz Q, Scott SM. Joint hypermobility and rectal evacuatory dysfunction: an etiological link in abnormal connective tissue? Neurogastroenterol Motil. 2010 Oct;22(10):1085-e283. doi: 10.1111/j.1365-2982.2010.01562.x. Epub 2010 Jul 5. PMID 20618831
- See also: Rome III Criteria — http://romecriteria.org